CLINICAL TRIAL: NCT03111082
Title: Incidence of Postoperative Neuromuscular Blockade in the Post-Anesthesia Care Unit at Parkland Hospital: Does Size Matter?
Brief Title: Incidence of Postoperative Neuromuscular Blockade in Post-Anesthesia Care Unit at Parkland Hospital: Does Size Matter?
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: STU 032017-054
Record Dates: First submitted 2017-04-07; First posted 2017-04-12 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Residual Neuromuscular Blockade
MeSH Terms: conditions — Delayed Emergence from Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Lean: BMI less than or equal to 29.9
- Obese: BMI between 30.0 and 39.9
- Morbidly Obese: BMI greater than or equal to 40.0

SUMMARY:
This prospective, observational study will assess 100 subjects in the post-anesthesia care unit (PACU) at Parkland Hospital. Upon arrival to the PACU, patients' train-of-four (TOF) ratio will be calculated using the StimPod NMS450 accelerometer to determine the presence of any residual paralysis. Any patient with a TOF ratio < 0.9 will be reassessed every 10 minutes until the ratio is ≥0.90. The time it takes to reach a TOF ratio ≥0.9 will be recorded. Subjects will be classified according to BMI categories: lean as <30 kg/m2, obese as 30≤BMI≤39.9 kg/m2, and morbidly obese as BMI ≥40 kg/m2. This data will serve as a baseline to assess the incidence of residual NMB that currently occurs in our PACU so that we may use this pilot data to design future studies that aim to reduce the incidence of residual NMB.

DETAILED DESCRIPTION:
Upon arrival to the PACU, patients enrolled in the study will be evaluated for residual paralysis with train-of-four (TOF) stimulation using the StimPod NMS450 accelerometer set to 30 mA. Any patients who have residual paralysis will be assessed Q10 minutes until the TOF ratio is ≥0.9. The time to achieve a TOF ratio ≥0.9 will be recorded. Any adverse events (e.g., hypoxia, reintubation, aspiration) that arise during the patient's PACU stay will be documented.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* Undergoing non-emergent surgery with general endotracheal anesthesia
* ASA physical status classification 1 to 4
* Willing and able to consent in English or Spanish
* No personal history of neuromuscular disease

Exclusion Criteria:

* Age less than 18 or older than 80
* Patient does not speak English or Spanish
* Planned postoperative intubation or ICU admission
* Allergy to sugammadex, neostigmine, glycopyrrolate, or rocuronium
* Family or personal history of malignant hyperthermia
* Patient refusal
* Monitored anesthesia care (MAC) or regional anesthesia planned
* Pregnant or nursing women
* "Stat" (emergent) cases
* Estimated creatinine clearance <30 mL/min
* Pre-existing muscle weakness of any etiology

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects in the post-anesthesia care unit who have undergone surgery with neuromuscular blockade
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2018-04-16 (Actual)

PRIMARY OUTCOMES:
Incidence of Residual Neuromuscular Blockade | 1 day on arrival to PACU
  To establish the current incidence of postoperative residual neuromuscular blockade (NMB), defined as a train-of-four ratio <0.9, in patients upon arrival to the PACU.

SECONDARY OUTCOMES:
Comparison of RNMB in Lean, Obese, and Morbidly Obese Patients | 1 day on arrival to PACU
  To assess the differences in the incidence of postoperative residual neuromuscular blockade (NMB) among PACU patients categorized based on body mass index (BMI) (lean, obese, and morbidly obese).

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Moon, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Health & Hospital System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No